CLINICAL TRIAL: NCT02541734
Title: Effect of Gelofusine on 111In-DTPA-AHX-Lys40-Exendin 4 Uptake in the Kidney
Brief Title: Effect of Gelofusine on GLP1-receptor Imaging
Acronym: GLP1-EX-GELO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL50233.091.14; 2014-003006-33 (EudraCT Number)
Record Dates: First submitted 2015-03-03; First posted 2015-09-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus
Keywords: SPECT; radiopeptides; gelofusine; Beta cell
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Polygeline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gelofusine and 111In-exendin 4 SPECT/CT (Experimental): subjects will receive a gelofusine injection before the injection of the radiopharmaceutical (111In-exendin 4)
  Interventions: Drug: Gelofusine; Radiation: 111In-exendin 4 SPECT/CT
- saline and 111In-exendin 4 SPECT/CT (Placebo Comparator): As a control, subjects will receive an injection of saline before the injection of the radiopharmaceutical (111In-exendin 4)
  Interventions: Radiation: 111In-exendin 4 SPECT/CT; Drug: Placebo

INTERVENTIONS:
Drug: Gelofusine — Infusion of gelofusine
  Arms: gelofusine and 111In-exendin 4 SPECT/CT
Radiation: 111In-exendin 4 SPECT/CT — 111In-exendin 4 SPECT/CT
Drug: Placebo
  Arms: saline and 111In-exendin 4 SPECT/CT

SUMMARY:
The highly promising and innovative tracer on 111In-DTPA-AHX-Lys40-Exendin 4 has been applied to determine beta cell mass in healthy volunteers and patients with type 1 diabetes. However, the high retention of the tracer in the kidneys was leading to a kidney/pancreas uptake ratio of 41±23. This high renal uptake is complicating absolute BCM quantification by SPECT imaging. In order to reduce the kidney/pancreas uptake ratio, investigators propose a co-infusion with the plasma expander Gelofusine since it has been shown in several pre-clinical and clinical studies that Gelofusine can reduce the renal retention of several other, closely related tracers. When investigators are able to reduce the kidney/pancreas uptake ratio, these findings will improve the interpretation of clinical quantitative SPECT, having important implications for therapeutic decision making for patients with diabetes, insulinomas or congenital hyperinsulinism, and may also have a major impact on our understanding of the pathophysiology of these diseases.

DETAILED DESCRIPTION:
Beta-cell imaging in vivo

Reliable, sensitive and specific non-invasive methods for comprehensive structural and functional characterization of living pancreatic beta-cells in vivo (and in vitro) would not only enhance our understanding of the pathophysiology of various diseases, but also enable longitudinal in vivo assessment of beta cell mass (BCM) and distribution in patients with e.g. diabetes (including patients who received beta cell replacement therapy). Additionally, it can help in diagnosing insulinomas and congenital hyperinsulinism and when coupled to other biomarkers it could aid patient stratification and enable patient-specific optimized treatment strategies.

Inhibiting the reabsorption of radiolabelled peptides

It has been shown, both in vitro and in vivo, that the kidney uptake of radiolabelled peptides can be reduced by co-infusion of agents that inhibit the reabsorption of these peptides. One of these agents is succinylated gelatin (Gelofusine), a plasma expander that consists of a mixture of collagen-derived peptides. Previous clinical observations have shown that Gelofusine infusion results in tubular proteinuria of both albumin and β2-microglobulin. Although the exact mechanism for this proteinuria is not completely understood, the megalin receptor system is most likely involved. Based on pre-clinical studies in mice and rats, it has been known that kidney uptake is significantly reduced for various tracers when co-infused with Gelofusine, like 111In-Octreotide 111In-Minigastrin, 68Ga-exendin-4 and 111In-DTPA-AHX-Lys40-Exendin 4. Additionally, it was shown that Gelofusine also reduces the renal retention of 111In- Octreotide by 45% in humans. In the current study, investigators will determine whether Gelofusine has also an effect on kidney retention of 111In-DTPA-AHX-Lys40-Exendin 4 in humans.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years
* <= 60 years
* Normal renal function
* Normal glucose regulation
* BMI 17>30

Exclusion Criteria:

* Use of any medication affecting renal function
* Known hypersensitivity to one of the substances used
* Hypertension
* Oedema
* Hypervolaemia
* Heart failure
* Pregnancy or the wish to become pregnant within 3 months after participation of the study.
* Lactation
* History of anaphylaxis
* Liver disease defined as aspartate aminotransferase or alanine aminotransferase level more than 3 times the upper limit of normal range (45U/L)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Renal uptake as measured by uptake of 111In-exendin-4 on SPECT images and without co-infusion of Gelofusine. | up to 8 months

SECONDARY OUTCOMES:
Pancreas uptake as measured by uptake of 111In-exendin-4 on SPECT images | up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gotthardt, Prof Dr, Principal Investigator — Radboud University Medical Center